CLINICAL TRIAL: NCT02261935
Title: Clustered, Randomized, Controlled Trial of the Home Care Nurse Carer Support Needs Assessment Practice Tool With Family Caregivers of Palliative Patients at Home
Brief Title: Supporting Family Caregivers of Palliative Patients at Home: the Carer Support Needs Assessment Intervention
Acronym: CSNAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kelli Stajduhar (Other)
Collaborators: Canadian Frailty Network (Other); Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor-Investigator, Kelli Stajduhar, Professor, University of Victoria
Organization: University of Victoria (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TVN-core2013-01 CCSRI-702597
Record Dates: First submitted 2014-09-30; First posted 2014-10-10 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Family Caregiving for a Palliative Patient
Keywords: Family caregiver; Home care nursing practice; Palliative care; End of life care; Family caregiver quality of life; Family caregiver grief symptoms; Family caregiver burden; Family caregiver preparedness for caregiving; Family caregiver perceived social supports; Family caregiver health status; Family caregiver satisfaction with healthcare provided

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Existing Home Care Nursing Practice (Active Comparator): Home care nurses provide care based on existing home care practice
  Interventions: Other: Existing home care nursing practice
- Practice Support Tool Intervention (Experimental): The practice support tool intervention will be the routine use of the Carer Support Needs Assessment Tool (CSNAT) in the practice of home care nurses (once every 4 weeks with each family caregiver) to document, monitor and address family caregiver support needs.
  Update - December 22, 2016 - In some home care offices only, a study nurse will meet with family caregivers who are in the intervention group to deliver the CSNAT intervention. Information arising from the CSNAT about family caregivers' support needs will be communicated by the study nurse to the home care nurse, and incorporated by the home care nurse into the home care plan for the patient and patient's family.
  Interventions: Other: Practice support tool intervention

INTERVENTIONS:
Other: Existing home care nursing practice — Home care nurses in this comparator group will provide "care as per usual" to their patients and family caregivers. The family is seen as the unit of care but no formal assessment of the caregiver will be done.
  Arms: Existing Home Care Nursing Practice
Other: Practice support tool intervention — The intervention will be the routine use of the Carer Support Needs Assessment Tool (CSNAT) in the practice of home care nurses (once every 4 weeks with each family caregiver) to document, monitor and address family caregiver support needs.
  The completed CSNAT tool will be kept in the patient chart and will be integrated into the care provided by the nurse.
  Update - December 22, 2016 - In some offices only, the CSNAT will be administered by a separate study nurse. Findings will be communicated to the home care nurse to inform the documenting, monitoring and addressing of family caregiver support needs.
  Other Names: CSNAT
  Arms: Practice Support Tool Intervention

SUMMARY:
In this project the investigators will train home care nurses to use the Carer Support Needs Assessment Tool (CSNAT) with a group of family caregivers (intervention group) and then compare the family caregivers' quality of life, burden and other outcomes to a group of family caregivers whose home care nurse is not using the CSNAT (control group). Findings will allow us to determine the effectiveness of using the CSNAT as a tool to identify, monitor and address family caregiver support needs in palliative home care.

DETAILED DESCRIPTION:
Caregiving places considerable burdens on family caregivers (FCG). While burden has been studied as a FCG outcome, it is also a predictor of other outcomes, including FCG quality of life (QoL). We have adapted a model of caregiver burden to hypothesize the various mechanisms by which addressing support needs may contribute to FCG QoL. In this model, support needs are closely associated with FCGs' perceived social support and preparedness for caregiving. These variables operate as (partial) mediators of the relationships between primary stressors, including patient functional dependence and symptom distress, and secondary appraisals, such as the perceived burden associated with caregiving, which, in turn influences FCGs QoL. The model further posits that FCGs' primary appraisal of patient caregiving needs (e.g., amount of care provided) is influenced by the functional dependence and symptom distress of the patient, and in turn influences perceived support, preparedness for caregiving, FCG burden, and, ultimately, FCG QoL. These variables are associated with a variety of demographic and health-related characteristics of the caregiver and patient.

Within the context of this conceptual framework outlined above, the CSNAT intervention is viewed as a mediator of the relationships between primary stressors and appraisals and FCG QoL (primary outcome). Also, the CSNAT intervention would lead to enhanced social support, preparedness, and reduced caregiver burden.

A clustered randomized control trial (RCT) design will be used to ascertain the effectiveness of the CSNAT as an intervention to improve the QoL of FCGs of patients receiving palliative care at home. Participating home care nurses will be randomized to one of two comparator groups (usual care and intervention) and the FCGs of their patients will be assigned to the corresponding comparator group. Data will additionally be collected over the same time frame and in the same manner from a non-randomized comparison usual care comparator group from a separate home care site where no nurses will be delivering the intervention, to help interpret the results (e.g., to determine the extent to which contamination may be have occurred). Update - August 31, 2015 - Due to low recruitment the non-randomized, comparison, usual care, comparator group has been discontinued.

Update - December 22, 2016 - Due to home care workloads of participant nurses and home care visit schedules in some participating home care offices, delivery of the intervention will be done by a dedicated study nurse (in some offices only). In these offices, family caregivers will continue to be assigned based on the randomized group assignment of their home care nurse. The dedicated study nurse will meet separately with FCGs who are in the intervention group to deliver the CSNAT intervention. Information arising from the CSNAT about family caregivers' support needs will be communicated by the study nurse to the home care nurse so that the home care nurse can incorporate this into the home care plan for the patient and patient's family. In home care offices that are not part of this change in procedures, the home care nurses in the intervention group will continue to deliver the CSNAT intervention during home care visits as before.

Our specific hypotheses are as follows:

* Hypothesis 1: The use of the CSNAT as a practice support tool intervention will lead to improved FCG QoL during the time prior to the patients' death and in bereavement.
* Hypothesis 2: The use of the CSNAT as a practice support tool intervention will contribute to the following secondary outcomes in FCGs during the time prior to the patient's death: enhanced perceived social support, improved preparedness to provide care and reduced caregiving burden.
* Hypothesis 3: CSNAT use during home care of patient before death will reduce grief symptoms during bereavement, among FCGs.

In addition to the RCT, qualitative and quantitative research will be conducted to understand the process related to implementing the CSNAT intervention in palliative home care and to explain the treatment results. We will specifically address the following questions:

* How are the CSNAT support needs being documented and met by home care nurses?
* How do home care nurses experience the use of the CSNAT in their daily practice?
* How comfortable are FCGs speaking to home care nurses about their own personal needs?
* To what extent are the relationships in the hypothesized conceptual framework supported?
* What is the relative importance of different CSNAT support needs with respect to FCG QoL and health during the illness trajectory, and the presence of post-bereavement grief symptoms?

ELIGIBILITY:
Inclusion Criteria:

For home care nurse participants:

* registered or licensed home care nurse at one of the following Vancouver Island Health Authority Home and Community Care offices: Victoria, Esquimalt/Westshore, Peninsula, Royal Oak, Duncan/Ladysmith, Oceanside, Comox Valley, Campbell River
* practiced in home care for > 6 months
* work a minimum of 10 shifts per month
* communicate well in English

For family caregiver participants:

* currently a family caregiver of palliative patient at home
* patient and family caregiver must be 18 years of age or older
* must communicate well in English

Exclusion Criteria:

For family caregiver participants

* diagnosed cognitive impairment
* identified safety risks in the home care environment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Trajectory of change in family caregiver quality of life while caring for a palliative patient at home, as measured by the Quality of Life in Life Threatening Illness - Family carer version (QOLLTI-F) total score | Baseline, 8 week intervals up to 96 weeks or patient death (whichever comes first)
  The QOLLTI-F is a self-report measure of family caregiver quality of life. It is composed of 16 items which assess the following 7 domains: state of carer, patient well-being, quality of care, outlook, environment, finances and relationships. Additional exploratory analyses will also be conducted on these subscales.
Family caregiver grief symptoms after patient death, as measured by the Texas Revised Inventory of Grief (TRIG) subscale scores | 12 weeks after patient death (will not be collected if patient death does not occur within the first 92 weeks of the study)
  The TRIG is a 21 item scale designed to assess grief symptoms. It relates to two points of time: past (immediate of shortly after the death) and present (the time of data collection). The 2 subscales measure a) feelings and actions at the time of the death and b) present feelings.

SECONDARY OUTCOMES:
Family caregiver quality of life after patient death, as measured by the Quality of Life in Life Threatening Illness - Family carer version Global Single-Item Scale (QOLLTI-F SIS) | 12 weeks after patient death
  The QOLLTI-F is a self-report measure of family caregiver quality of life. We will be using the score from the single item score measuring global quality of life (Part A).
Trajectory of change in family caregiver burden while caring for a palliative patient at home, as measured by the Family Appraisal of Caregiving Questionnaire for Palliative Care (FACQ-PC) Scale | Baseline, 8 week intervals up to 96 weeks or patient death (whichever comes first)
  A 25 item measure of family caregiver's positive and negative appraisals of caregiving, including strain, positive appraisals, distress, and family wellbeing.
Trajectory of change in family caregiver preparedness for caregiving while caring for a palliative patient at home, as measured by the Family Caregiving Inventory: Preparedness Scale | Baseline, 8 week intervals up to 96 weeks or patient death (whichever comes first)
  A caregiver self-rated instrument that consists of 8 items that asks caregivers how well prepared they believe they are for multiple domains of caregiving. Preparedness is defined as perceived readiness for multiple domains of the caregiving role such as providing physical care, providing emotional support, setting up in-home support services, and dealing with the stress of caregiving.
Trajectory of change in family caregiver perceived social supports while caring for a palliative patient at home, as measured by the Medical Outcome Survey (MOS) Social Support Survey | Baseline, 8 week intervals up to 96 weeks or patient death (whichever comes first)
  Overall Support Index determined using the mean from 18 items within four sub-measures and the mean from the additional item; (a) emotional/information support, (b) tangible support, (c) affectionate support, and (d) positive social interaction support. Designed to assess the perceived availability of social support.
Trajectory of change in family caregiver health status and mental health status while caring for a palliative patient at home, as measured by the Veterans RAND 12 item health survey | Baseline, 8 week intervals up to 96 weeks or patient death (whichever comes first)
  A 14 item scale, 12 of which are a sampling of items from each of the eight domains of health (physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems and mental health). The eight scales are summarized into two summary scores, physical (PCS) and mental (MCS).
Trajectory of change in family caregiver satisfaction with healthcare provided while caring for a palliative patient at home until death, as measured by the Canadian Health Care Evaluation Project - Caregiver Questionnaire (CANHELP LITE) | Baseline, 8 week intervals up to 96 weeks or patient death (whichever comes first), 12 weeks after patient death (will not be collected if patient death does not occur within the first 92 weeks of the study)
  Overall score calculated as the unweighted average of all 21 items (22 for the bereavement version which will be used after patient death) answered. A tool to evaluate satisfaction with care for family members of older patients with life threatening illnesses up to and until death.

CONTACTS AND LOCATIONS:
Overall Officials: Kelli I Stajduhar, PhD, Principal Investigator — University of Victoria; Richard G Sawatzky, PhD, Principal Investigator — Trinity Western University
Locations (1):
- Vancouver Island Health Home and Community Care, Victoria, British Columbia, Canada

REFERENCES:
- [Derived] Ryan RE, Connolly M, Bradford NK, Henderson S, Herbert A, Schonfeld L, Young J, Bothroyd JI, Henderson A. Interventions for interpersonal communication about end of life care between health practitioners and affected people. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD013116. doi: 10.1002/14651858.CD013116.pub2. PMID 35802350